CLINICAL TRIAL: NCT06398366
Title: Cardiac Abnormalities in Stroke Prevention and Risk of Recurrence (CASPR): a Multi-center Observational Cohort Study
Brief Title: Cardiac Abnormalities in Stroke Prevention and Risk of Recurrence
Acronym: CASPR
Status: Enrolling by invitation | Type: Observational
Sponsor: The Cooper Health System (Other)
Collaborators: Duke University (Other); Covenant Health, Canada (Other); University of Colorado, Denver (Other); Medical University of South Carolina (Other); University of Maryland, Baltimore (Other); University of Pennsylvania (Other); Emory University (Other); University of Chicago (Other); University of Tennessee (Other); Ohio State University (Other); West Virginia University (Other); Mayo Clinic (Other); Boston Medical Center (Other); Rhode Island Hospital (Other); Beth Israel Lahey Health (Unknown); Christiana Care Health Services (Other); Henry Ford Health System (Other); Thomas Jefferson University (Other); University of Iowa (Other); University of California, Los Angeles (Other); Allina Health System (Other); Yale University (Other); The University of Texas Health Science Center, Houston (Other); Dartmouth-Hitchcock Medical Center (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Jesse Thon, Principal Investigator, The Cooper Health System
Other Study IDs: 22-165
Record Dates: First submitted 2023-12-14; First posted 2024-05-03 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cryptogenic Stroke
Keywords: carotid atherosclerosis; heart failure; cardiomyopathy; embolic stroke
MeSH Terms: conditions — Ischemic Stroke; Carotid Artery Diseases; Heart Failure; Cardiomyopathies; Embolic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cooper Health System: Patients from Cooper Health System and additional sites

SUMMARY:
This is a multi-center retrospective analysis of consecutive adult patients with cryptogenic stroke patients following a comprehensive workup for the underlying stroke etiology. Patients will be eligible for inclusion if the index stroke event occurred between 1/1/2016 and 06/30/2022.

DETAILED DESCRIPTION:
This is an exploratory observational cohort study of existing registry-based clinical, laboratory, and radiographic data. There are multiple pre-specified hypotheses that will be tested using this data set, which include the entire cohort as well as planned subgroup analyses. The analyses center around patients with cryptogenic stroke (no clear stroke mechanism) but who are characterized by "potential embolic sources". These include but are not limited to: left atrial enlargement or dysfunction, left ventricular dysfunction /heart failure with reduced ejection fraction (HFrEF), patent foramen ovale (PFO), paroxysmal atrial fibrillation (pAF), lambl's excrescence, valvular lesions, carotid web, and nonstenotic cervical arterial plaque. A brief summary of several planned hypothesis is itemized below:

1. To evaluate treatment practices in patients with potential embolic sources.
2. To estimate the risk of recurrent stroke, major bleeding, and/or death following an incident stroke event across various potential embolic sources.
3. To compare rates of recurrent stroke, major bleeding, and/or death across various potential embolic sources, when stratified by antithrombotic treatment type.
4. To evaluate type, frequency, and findings of long-term outpatient cardiac event monitoring (for paroxysmal atrial fibrillation). And furthermore, to determine antithrombotic treatment changes following abnormalities detected with such monitoring.
5. To develop and validate a risk prediction model for later atrial fibrillation in cryptogenic stroke by integrating a machine-learning algorithm or convolutional neural network analysis of 12-lead electrocardiographic data with clinical, laboratory, and radiographic parameters.
6. To develop and validate a risk prediction model for later atrial fibrillation, atrial fibrillation burden, and recurrent stroke and/or death using a machine-learning and/or convolutional neural network and/or validated electrophysiologic biomarkers (e.g., p-wave morphology) abstracted from outpatient telemetry, when added to clinical and radiological patient profiles.
7. To compare the sensitivity of various outpatient cardiac telemetry devices for identifying atrial fibrillation.
8. To evaluate real-world treatment practices of patent foramen ovale closure, antithrombotic therapy in patent foramen ovale, and risk of stroke recurrence.
9. To evaluate real-world secondary stroke prevention strategies in patients with heart failure, with and without left ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive adult patients (18 yrs of age or older) diagnosed with cryptogenic stroke despite complete neurodiagnostic workup, including the following:

   A. Transthoracic echocardiogram B. EKG and 24h minimum cardiac telemetry C. Cervical and intracranial vessel imaging D. No known and established source of cerebral embolism after completion of the aforementioned testing E. CT or MRI evidence of acute cerebral infarction F. Onset of stroke or last known well within 2 weeks of hospitalization or study inclusion start date (unless time last known well is unknown)
2. Left ventricular ejection fraction greater than or equal to 20%

Exclusion Criteria:

1. Patients with an established stroke mechanism that is diagnosed prior to or at the time of the index stroke event. Examples include but are not limited to:

   A. New diagnosis of atrial fibrillation during index stroke admission, or history of prior atrial fibrillation B. Cervical or intracranial atherosclerosis in a vessel supplying the infarcted brain region, with 50% luminal stenosis by NASCET criteria C. Cervical or intracranial arterial dissection D. Inflammatory vasculopathy (e.g., giant cell arteritis, primary central nervous system angiitis) E. Acute myocardial infarction or cardiac arrest at the time of stroke F. Intracardiac thrombus (e.g., left ventricular, left atrial, left atrial appendage thrombus), irrespective of cardiac function G. Small vessel disease (defined by the presence of a single, subcortical infarction less than 1.5cm in diameter on computed tomography, less than 2.0cm in diameter on diffusion-weighted imaging, or without radiographic evidence of infarction BUT with symptoms consistent with a subcortical syndrome-e.g., pure motor hemiparesis, pure hemisensory impairment, mixed motor-sensory syndrome, ataxic hemiparesis, or dysarthria-clumsy hand syndrome)
2. Patients without follow-up information at 30 days (although patients who expired within 90 days of stroke are still eligible for inclusion)
3. Patients enrolled in a randomized clinical trial in which antithrombotic group is blinded to the investigator
4. Transient ischemic attack
5. Primary intracerebral hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (18 yrs of age or older) diagnosed with cryptogenic stroke despite complete neurodiagnostic workup. Patients admitted between 1/1/2016 and 6/30/2022 with acute ischemic stroke will be screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of potential embolic sources | through study completion, an average of 2 years
  Epidemiological estimates of prevalence of various potential embolic sources in the cryptogenic stroke population will be calculated across the cohort
The odds of recurrent stroke, major bleeding (according to the International Society of Thrombosis and Hemostasis), and/or death will be estimated across the cohort, with annualized event rates also calculated | At any point during follow-up over a minimum of 90 days after stroke (average of 2 years)
  . This outcome will be evaluated across each subgroup of potential embolic source (e.g., valvular lesions present vs. absent, nonstenotic carotid plaque present or absent). Adjusted estimates of event probability will be calculated between patients treated with various antithrombotic types (or class, e.g. anticoagulant vs. antiplatelet) using propensity score matching according to propensity of antithrombotic use
Number of patients treated with antiplatelet, anticoagulant, or combination antithrombotic therapy | through study completion, an average of 2 years
  Following the index cryptogenic stroke, the outcome of specific antithrombotic treatment will be compared between patient groups (antiplatelet, anticoagulant, combination antithrombotic)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Thon, Principal Investigator — Cooper Health System
Locations (1):
- Cooper Health System, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegler JE, Goicoechea EB, Penckofer M, Eklund K, Yaghi S, Stretz C, Lineback CM, Stamm B, Peter S, D'Souza M, Conyers FG, Khasiyev F, Kerrigan D, Lewis S, Ali H, Aboul-Nour H, Sharma R, Nahab FB, Glover P, Thompson SL, Alshaer QN, Thottempudi N, de Havenon A, Culbertson CJ, Melkumova E, Chionatos RA, Jillella DV, Daniel JA, Ro J, Frankel MR, Dumitrascu OM, Brown S, Parikh P, Doolittle C, Yahnke I, Sathya A, Kang J, Kirchhoffer K, Bowman A, Smith MM, Brorson JR, Asabere A, Shahrivari M, Elangovan C, Sheibani N, Krishnaiah B, Gaudio E, Sloane KL, Rothstein A, Alvi MM, Annam S, Amankwah C, Kam W, Abburi N, Farooqui M, Rojas-Soto D, Molaie A, Khezri N, Zubair AS, Abbasi M, Van Coevering RJ, Chen L, Nedelcu S, Herpich F, Chahien D, Sehgal S, Liebeskind DS, Linares G, Zha A, Sarkar M, Xi R, Nelson A, Abu Qdais A, Al Kasab S, Singh E, Patel V, Aziz YN, Mehndiratta P, DeMarco A, Sharrief A, Cucchiara B, Salehi Omran S, Nguyen TN, Dubinski M, Ackerman J, Thon J. Outcomes of Patients With Embolic Stroke of Undetermined Source Treated With Antiplatelet Agents or Anticoagulation: A Multicenter Cohort Study. Neurology. 2025 Aug 12;105(3):e213876. doi: 10.1212/WNL.0000000000213876. Epub 2025 Jul 3. PMID 40609061